CLINICAL TRIAL: NCT06346951
Title: Survey on the Current Status of IFD Diagnosis and Treatment by Intensive Care Physicians in Sichuan Province (IFS)
Acronym: IFS
Status: Not yet recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lingai Pan, Associate Clinical Professor, Sichuan Provincial People's Hospital
Other Study IDs: LPan
Record Dates: First submitted 2024-03-07; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this survey is to learn about the current status of the diagnosis and treatment of invasive fungal infections among intensive care physicians in Sichuan Province (IFS). Its primary focus lies on answering the following questions: ①awareness and proficiency in diagnosis and treatment; ②the use of antifungal medications; ③the application of microbiological identification and diagnostic methods. We aim to analyze the problems and deficiencies that existed among intensive care physicians in order to provide a basis for the development of targeted training and intervention measures.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care physicians in medical institutions at all levels in Sichuan Province

Exclusion Criteria:

* Exclude non-Sichuan physicians.
* Excluding physicians who are not engaged in intensive care unit.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Intensive care physicians in medical institutions at all levels in Sichuan Province. Anticipated total of 20 centers will participate in the study, with a total of 300 physicians to be included in the survey.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The survey on the hospital's diagnostic and treatment standards and infrastructure for invasive fungal infections | From enrollment to the end of survey at 16 weeks
  ①To investigate the basic knowledge and skill mastery of invasive fungi diagnosis and treatment by intensive care physicians in Sichuan province, including information on pathogenesis, clinical manifestations, diagnosis, and treatment.
  ② To investigate the concerns and selection tendency of intensive care physicians in Sichuan province in choosing antifungal drugs in practice, including information on treatment types, drug choice, dosage, and treatment course.
The survey on the awareness of an invasive fungal infection among intensive care physicians | From enrollment to the end of survey at 16 weeks
  ① To assess the application of pathogenetic detection and diagnostic methods of invasive fungal infections by intensive care physicians in Sichuan Province, including the technical level of fungal smear and culture, PCR detection, histopathological examination, and NGS.
  ②To analyse the problems and deficiencies in the diagnosis and treatment of invasive fungal infections among invasive care physicians in Sichuan Province, and to provide a reference basis for the development of targeted training and intervention measures.

IPD SHARING:
Plan to Share IPD: Undecided